CLINICAL TRIAL: NCT07406087
Title: Adaptation and Implementation of an Evidence-Based Patient Navigation Intervention for Adolescent and Young Adult Cancer Survivors
Brief Title: Navigation Intervention for Adolescent and Young Adult Cancer Survivors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UG3CA297705 (NIH); 1UG3CA297705-01A1 (NIH)
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Ovarian Cancer; Cervical Cancer; Testicular Cancer; Colon Rectal Cancer; Melanoma (Skin Cancer); Endometrial Cancer; Sarcoma; Thyroid Cancer
Keywords: Adolescent and Young Adult; Cancer Survivors; Patient Navigation; Adaptations; Implementation Science
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Testicular Neoplasms; Colonic Neoplasms; Melanoma; Endometrial Neoplasms; Sarcoma; Thyroid Neoplasms

STUDY DESIGN:
Intervention Model Description: After input from focus groups, we will conduct a prospective, single-arm pilot study of the adapted navigation program and refine the program to enhance acceptability to patients and clinicians, enhance feasibility and effectiveness, and develop and pilot pragmatic trial evaluation tools and methods prior to the start of the UH3 phase of the trial, which will be a pragmatic stepped wedge prospective trial. Objectives will be updated for the UH3 phase once awarded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adapted Patient Navigation Program (Experimental): The primary objectives in the UG3 phase of the study are to adapt and tailor an existing patient navigation program to meet the needs of AYA cancer survivors and the local clinical context. Adolescent and young adult cancer survivors will be enrolled in a single arm pilot study of the adapted navigation program.
  Interventions: Other: Adapted patient navigation program targeting adolescent and young adult cancer survivors

INTERVENTIONS:
Other: Adapted patient navigation program targeting adolescent and young adult cancer survivors — In the UG3 phase, we will be adapting a patient navigation intervention to suit adolescent and young adult cancer survivors and conducting a single-site pilot test of the adapted intervention. We will conduct a pilot test of the adapted AYA PN program at a single participating site, focusing on the perceptual implementation outcomes of acceptability, appropriateness, and feasibility and the hypothesized patient navigation program outcomes of increased motivation, capability, and opportunity for care. The pilot will also include testing of the patient identification algorithm-which we have high confidence in and have used for other studies-patient enrollment/engagement methods, clinical workflow, survey recruitment methods, and health IT elements (e.g., access, ease of use).

SUMMARY:
We propose to: 1) Adapt an evidence-based cancer-focused patient navigation (PN) program for the Adolescent and Young Adult (AYA) cancer survivor population; and 2) Plan and conduct an effectiveness-implementation trial of this program within Kaiser Permanente Southern California (KPSC). PLEASE NOTE: This study is awarded in two phases. The UG3 phase has been awarded for the first two years; upon successful completion of this phase by meeting pre-defined milestones, the National Cancer Institute (NCI) will provide funding for the second phase of the study (Years 3-6), which will allow our team to conduct a trial to determine the effectiveness of the implementation of the adapted PN program for the AYA cancer survivor population. Here we are focused on the initial UG3 phase and will update the protocol for the UH3 trial upon successful completion of the UG3 milestones and receipt of the UH3 award.

The primary objectives in the UG3 phase of the study are to adapt and tailor an existing PN program to meet the needs of AYA cancer survivors and the local clinical context via (a) interviews with key stakeholders (patients, clinicians, administrators) and (b) guidance from our AYA Primary Care Survivorship Council. We will conduct a pilot study of the adapted PN program and refine the program to enhance acceptability to patients and clinicians, enhance feasibility and effectiveness, and develop and pilot evaluation tools and methods prior to the start of the UH3 phase of the trial, which will be a larger trial. Objectives will be updated for the UH3 phase once awarded.

DETAILED DESCRIPTION:
In the UG3 phase, we will be adapting a patient navigation (PN) intervention to suit adolescent and young adult (AYA) cancer survivors and conducting a single-site pilot test of the adapted intervention. In the UH3 phase, we will conduct a pragmatic stepped wedge hybrid effectiveness implementation trial evaluating (1) clinical effectiveness and (2) implementation outcomes, across a range of data sources.

Intervention:

Navigator-level: For the pilot test in the UG3 phase, we will provide PN training for the adapted AYA PN program to at least one navigator. We anticipate that navigators will undergo a comprehensive training curriculum that draws on existing Kaiser Permanente Southern California (KPSC) PN program trainings (e.g., KP Motivational Interviewing for Clinicians, KPSC Panel Management) and includes primary care and cancer survivorship/surveillance components and established recommendations for cancer survivorship navigation from the American Society of Clinical Oncology (ASCO) and others. These resources include core navigation competencies for survivorship, patient assessment, scope of practice, etc. These trainings will be completed with additional focus areas/domains identified during the adaptation processes. Based on the structure of the existing PN program, we anticipate holding monthly review of navigation milestones and metrics (developed based on established recommendations and stakeholder input) with the study team.

Patient-level: For the pilot test in the UG3 phase, we will identify eligible patients from a single clinical site within KPSC. We anticipate enrolling 15-25 patients in the pilot. Patients will receive a letter and brochure describing the adapted AYA PN program with a bio of their assigned navigator and how the program will help integrate primary care and cancer survivorship needs. We strongly anticipate navigation 'touches' will include progressive steps via a combination of delivery modes as with the existing PN programs: 1) email: patients with KP.org patient portal accounts will receive email communication from navigators; 2) text: patients with registered mobile phone in KP membership files will receive text-based communications; 3) calls: patients will receive calls from their navigator to discuss scheduling, overdue recommended care, and motivational coaching; 4) letters: patients may receive letters if unable to be reached via email, text, and calls. Navigators will work with the electronic medical record (EMR) to identify need for recommended healthcare services and gaps in care, working with the care team to pend orders for physician review and work directly with the patient using motivational interviewing skills to encourage participation in care, address social needs, and identify care goals. PN program milestones, developed based on established recommendations for survivorship navigation metrics and the input from our adaptation processes, will likely include patients contacted, engagement activities, and pending orders for physician review for overdue services.

System-level: As part of the UG3 phase, we will work closely with our partners to adapt the PN program to suit existing clinical needs and workflows. We will convene 2-3 focus groups with care teams (nurses/physicians/advanced practice providers) and department administrators (DAs) using a semi-structured focus group format. These groups will provide feedback on the team-based care focus for the PN program, how to integrate seamlessly into existing clinical workflows, suggestions for use and/or expansion of existing KPSC information technology (IT) tools (e.g., the Complete Care Model tools), and clinical needs of the patient population. Using adapted health IT tools, flags may be created for patients due for recommended services.

In the UG3 phase, the study will open enrollment for the prospective single-arm pilot study by month 18, after focus group data and program adaptation is complete. Completion of data collection for the pilot is estimated at month 24.

In the UG3 phase, the patients in the single site pilot will complete all study tasks by 6 months.

Following the structure of the NCI two-phase cooperative agreement, we propose to: 1) Adapt an existing evidence-based, cancer-focused PN program to the AYA survivor population and to the clinical setting; and 2) Conduct a pragmatic stepped wedge hybrid type 2 effectiveness-implementation trial within a large integrated healthcare system, Kaiser Permanente Southern California (KPSC). We hypothesize that the adapted PN program will lead to increased uptake of high-quality, guideline-recommended primary care and cancer surveillance services for AYA survivors (clinical outcomes), and high levels of acceptability, appropriateness, feasibility, adoption, penetration, fidelity, and sustainment. We have defined measurable, feasible milestones for both the UG and UH phases of the proposal.

In the UG3 phase, we will engage in a three-step process to achieve our goals:

1. Intervention refinement via context assessment including multilevel barriers and facilitators to guide adaptation; adaptation and tailoring to local contexts.
2. Demonstrate feasibility of program implementation with pilot testing of recruitment, data collection, evaluation plans and methods, and data sources.
3. Develop and demonstrate the feasibility of logistical and administrative arrangements for conducting the pragmatic trial in the UH3 phase including finalizing agreements with sites, IRB approvals, and development of a manual of operations for the trial.

In step 1, we plan for rigorous exploration and documentation of adaptation processes via a combined use of implementation and adaptation frameworks, representing a significant contribution to the field. Intentional adaptation provides an opportunity for implementation flexibility, potentially improving the overall fit of an evidence-based intervention to a new population and/or context (Kirk et. al, 2020), such as AYA survivors care in the primary care setting. Several adaptation frameworks have been proposed over the past decade, with a collective recognition of the importance of rigorous research on adaptation processes and the distinction between the function (e.g., core elements) and form (e.g., delivery type) of evidence-based interventions. (Chambers, 2023). We will follow the overarching steps of adaptation processes as described by Escoffery et al. (2019), consisting of eleven discrete steps, with extensive stakeholder engagement throughout. We will supplement this with a novel application of the RE-AIM framework for guidance on the 'who, why, how' of adaptation a nascent and exciting application of RE-AIM to adaptation processes. We will use the FRAME to guide thorough documentation of adaptation activities throughout the eleven steps. This blend of Escoffery's eleven steps, RE-AIM, and FRAME provides a stepwise, thoughtful approach for capturing the rationale for adaptation, the internal and external context of adaptation, and for cataloguing adaptation elements.

Recent work from leaders in the field have combined RE-AIM with adaptation frameworks (Rabin et. al, 2018; Cohen et. al, 2023), although not in this specific combination which is more appropriate to address our research questions. We propose a multilevel adaptation process, tailoring PN program components to meet the needs of AYA cancer survivors, primary care teams, and the organizational setting (and leveraging available supportive resources). We will be adapting KPSC's existing PN program for patients newly diagnosed with cancer, which includes KPSC's robust 'Complete Care' model and health IT tools shown to be effective at managing cancer (diagnosis and initial treatment) and other chronic conditions (Henry et. al, 2016; Kanter et. al, 2013). In step 2, we will conduct a pilot study of the adapted PN program with a single clinic, collecting patient, clinician, and clinic-level data and iteratively refining the PN program as appropriate. Lastly, in step 3 we will develop our trial manual of operations and obtain administrative and other approvals so that the trial is set to launch at start of Year 3.

In the UH3 phase, we will conduct a pragmatic stepped wedge hybrid type 2 effectiveness-implementation trial with extensive quantitative and qualitative process evaluation activities to examine mechanisms of effect, moderators and other contextual factors. This protocol will be updated once the UH3 phase is awarded.

ELIGIBILITY:
Inclusion Criteria:

* patients of current age of 21-45 years who received a diagnosis of breast, ovarian, cervical, testicular, colon/rectal, melanoma, endometrial, sarcoma, or thyroid cancer.

Exclusion Criteria:

* Exclusion criteria: patients with a history of leukemia or lymphoma; patients with metastatic disease at diagnosis; and patients with less than 120 days of Kaiser Permanente Southern California insurance membership after diagnosis of primary cancer.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-11-01 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Self-Efficacy Measurement | From enrollment to completion at 6 months post-enrollment
  Patient survey outcome
Measures of Care Coordination and Communication Measurement | From enrollment to completion at 6 months post-enrollment
  Patient Survey Outcome
Barriers to Care Measurement | From enrollment to 6 months post-enrollment
  Patient Survey Outcome
Appropriateness/Acceptability of the Program Measurement | From enrollment to completion at 6 months post-enrollment
  Patient Survey Outcome
Integration of the Navigation Program Measurement | Patient enrollment to 6 months post-patient enrollment
  Clinician/Administrator Survey Outcome
Appropriateness/Acceptability Measurement | Patient enrollment to 6 months post-patient enrollment
  Clinician/Administrator Survey Outcome
Feasibility Measurement | Patient enrollment to 6 months post-enrollment
  Clinician/Administrator Survey Outcome

CONTACTS AND LOCATIONS:
Overall Officials: Erin E Hahn, PhD, Principal Investigator — Kaiser Permanente Southern California, Department of Research & Evaluation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nekhlyudov L, O'Malley D M, Hudson SV. Integrating primary care providers in the care of cancer survivors: gaps in evidence and future opportunities. Lancet Oncol. Jan 2017;18(1):e30-e38. doi:10.1016/S1470-2045(16)30570-8
- [Background] McCabe MS, Partridge AH, Grunfeld E, Hudson MM. Risk-based health care, the cancer survivor, the oncologist, and the primary care physician. Seminars in oncology. Dec 2013;40(6):804-12. doi:10.1053/j.seminoncol.2013.09.004
- [Background] DiMartino L LP, Mittman B. Increasing the quantity and quality of coordinating center activity in implementation science: A novel application of core function/form concepts. . presented at: Paper accepted at 16th Annual Conference on the Science of Dissemination and implementation; December 10-13, 2023 Washington, DC;.
- [Background] Lengnick-Hall R, Stadnick NA, Dickson KS, Moullin JC, Aarons GA. Forms and functions of bridging factors: specifying the dynamic links between outer and inner contexts during implementation and sustainment. Implementation Science. 2021/04/01 2021;16(1):34. doi:10.1186/s13012-021-01099-y
- [Background] Esmail LC, Barasky R, Mittman BS, Hickam DH. Improving Comparative Effectiveness Research of Complex Health Interventions: Standards from the Patient-Centered Outcomes Research Institute (PCORI). J Gen Intern Med. Nov 2020;35(Suppl 2):875-881. doi:10.1007/s11606-020-06093-6
- [Background] Perez Jolles M, Lengnick-Hall R, Mittman BS. Core Functions and Forms of Complex Health Interventions: a Patient-Centered Medical Home Illustration. J Gen Intern Med. Jun 2019;34(6):1032-1038. doi:10.1007/s11606-018- 4818-7
- [Background] Khor S HP, Basu A, Haupt EC, Lyons LJ, Hahn EE, Bansal A. Racial Disparities in the Ascertainment of Cancer Recurrence in Electronic Health Records. JCO Clinical Cancer Informatics. 2023;e2300004
- [Background] Hahn EE M-PC, Pounds D, Lyons LJ, Lee JS, Shen E, Hong BD, La Cava S, Brasfield FM, Durna LN, Kwan KW. Effect of a community-based medical oncology depression screening program on behavioral health referrals among patients with breast cancer: a randomized clinical trial. JAMA 2022;327(1):41-49.
- [Background] Xie F, Lee J, Munoz-Plaza CE, Hahn EE, Chen W. Application of Text Information Extraction System for Real-Time Cancer Case Identification in an Integrated Healthcare Organization. J Pathol Inform. 2017;8:48. doi:10.4103. https://doi.org/10.4103/jpi.jpi_55_17
- [Background] Cook AJ, Delong E, Murray DM, Vollmer WM, Heagerty PJ. Statistical lessons learned for designing cluster randomized pragmatic clinical trials from the NIH Health Care Systems Collaboratory Biostatistics and Design Core. Clin Trials. Oct 2016;13(5):504-12. doi:10.1177/1740774516646578
- [Background] NIH Pragmatic Trials Collaboratory. Rethinking Clinical Trials: A Living Textbook of Pragmatic Clinical Trials. Accessed on 1/30/2024: https://rethinkingclinicaltrials.org/.
- [Background] 107. Tuzzio L, Larson EB. The Promise of Pragmatic Clinical Trials Embedded in Learning Health Systems. EGEMS (Wash DC). Apr 3 2019;7(1):10. doi:10.5334/egems.285
- [Background] Kirsty L, Shaun T, Frank S, Peter D, Kevin ET, Merrick Z. The PRECIS-2 tool: designing trials that are fit for purpose. BMJ : British Medical Journal. 2015;350:h2147. doi:10.1136/bmj.h2147
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Medical care. 2012;50(3):217-226. doi:10.1097/MLR.0b013e3182408812
- [Background] Kanter MH LG, Bellows J, Chase A. Complete care at Kaiser Permanente: transforming chronic and preventive care. The Joint Commission Journal on Quality and Patient Safety. 2013;39(11):484-94.
- [Background] Henry SL, Shen E, Ahuja A, Gould MK, Kanter MH. The Online Personal Action Plan: A Tool to Transform Patient- Enabled Preventive and Chronic Care. American journal of preventive medicine. Jul 2016;51(1):71-7. doi:10.1016/j.amepre.2015.11.014
- [Background] Cohen AJ, Russell LE, Elwy AR, et al. Adaptation of a social risk screening and referral initiative across clinical populations, settings, and contexts in the Department of Veterans Affairs Health System. Original Research. Frontiers in Health Services. 2023;2
- [Background] Rabin BA, McCreight M, Battaglia C, et al. Systematic, Multimethod Assessment of Adaptations Across Four Diverse Health Systems Interventions. Methods. Frontiers in Public Health. 2018;6
- [Background] Escoffery C, Lebow-Skelley E, Udelson H, Böing EA, Wood R, Fernandez ME, Mullen PD. A scoping study of frameworks for adapting public health evidence-based interventions. Transl Behav Med. Jan 1 2019;9(1):1-10. doi:10.1093/tbm/ibx067
- [Background] Chambers DA. Advancing adaptation of evidence-based interventions through implementation science: progress and opportunities. Perspective. Frontiers in Health Services. 2023;3
- [Background] Kirk MA, Moore JE, Wiltsey Stirman S, Birken SA. Towards a comprehensive model for understanding adaptations' impact: the model for adaptation design and impact (MADI). Implementation Science. 2020/07/20 2020;15(1):56. doi:10.1186/s13012-020-01021-y

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2026-01-27): https://cdn.clinicaltrials.gov/large-docs/87/NCT07406087/Prot_SAP_000.pdf